CLINICAL TRIAL: NCT00526435
Title: Evaluation of the Walk With Ease Program Among People With Arthritis
Brief Title: Evaluation of Walk With Ease in Arthritis
Acronym: WWE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina, Chapel Hill (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-AAMC-0975; AAMC-0975
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Arthritis
Keywords: Arthritis; osteoarthritis; rheumatoid arthritis; fibromyalgia; lupus
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Fibromyalgia | interventions — Walking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group WWE (Experimental): Subjects will participate in a group-assisted 6 week WWE program.
  Interventions: Behavioral: Walk with Ease - Group
- Self-directed (Experimental): Subjects will follow the self-directed WWE program.
  Interventions: Behavioral: Walk with Ease - Self

INTERVENTIONS:
Behavioral: Walk with Ease - Group — Participate in 6-week, 1 hour per week group assisted classes (with instructor).
  Arms: Group WWE
Behavioral: Walk with Ease - Self — SUbject will receive the WWE workbook and follow it without group/instructor assistance.
  Arms: Self-directed

SUMMARY:
The overall goal of this study is to determine the whether the Walk with Ease (WWE) program in its 2 version (group-assisted and self-directed) can increase physical activity and fitness levels among individuals (18 years and older) with arthritis over the long-term. Participants will be approximately 657 subjects from 20-24 rural and urban communities across North Carolina. It is expected that participants in the WWE program will have reduced pain, improved function and increased activity levels after participation in this 6-week program.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported, doctor-diagnosed arthritis
* Ages 18+

Exclusion Criteria:

* Non-English speaking
* Severe impairment of physical or mental function
* Co-existing condition for which exercise is contraindicated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | 6 weeks
6-minute walk | 6 weeks
Walking behaviors | 6 weeks
Exercise self-efficacy | 6 weeks

SECONDARY OUTCOMES:
Health-related Quality of Life (SF36)
Health Assessment Questionnaire
Arthritis Symptoms
Senior Fitness Test (function)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hootman, PhD, Study Director — Centers for Disease Control and Prevention; Leigh F Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States